CLINICAL TRIAL: NCT05325853
Title: A Randomized, Single-Masked, Active-Controlled, Parallel-Group Evaluation of Safety and the Local Anesthetic Effect of Articaine Sterile Topical Ophthalmic Solution (AG-920) in a Pediatric Population
Brief Title: A Study of Safety and the Local Anesthetic Effect of AG-920 Ophthalmic Solution in a Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Genomics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AG-920-CS304
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia, Local
Keywords: AG-920; Articaine; Septocaine; Intravitreal Injection; Proparacaine
MeSH Terms: interventions — Carticaine; proxymetacaine

STUDY DESIGN:
Intervention Model Description: Subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive a single dose of AG-920 or proparacaine into one (study) eye (2 drops 30 seconds apart).
Who Masked: Participant
Masking Description: The study is single masked. Treatment assignments will be masked to the subjects and their parent/legal guardian only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG-920 (Experimental): Articaine Sterile Topical Ophthalmic Solution (AG-920) is a sterile, isotonic, non-preserved aqueous solution containing the active ingredient Articaine HCl 8%.
  Interventions: Drug: AG-920
- Proparacaine (Active Comparator): 0.5% Proparacaine Hydrochloride
  Interventions: Drug: Proparacaine Ophthalmic

INTERVENTIONS:
Drug: AG-920 — AG-920 Sterile Topical Ophthalmic Solution
  Other Names: articaine
  Arms: AG-920
Drug: Proparacaine Ophthalmic — 0.5% Proparacaine Hydrochloride
  Other Names: Proparacaine
  Arms: Proparacaine

SUMMARY:
A Phase 3, randomized, active-controlled, study in pediatric subjects. It is designed to evaluate the safety and anesthetic efficacy of one dose of AG-920 ophthalmic solution compared to Proparacaine Hydrochloride Ophthalmic Solution.

DETAILED DESCRIPTION:
A Phase 3, randomized, active-controlled, single-masked, parallel-group design study in pediatric subjects performed in the US. It is designed to evaluate the safety and anesthetic efficacy of one dose of AG-920 compared to Proparacaine. In this study, parent/legal guardians will provide informed consent (and where applicable, subjects will provide assent). Subjects who fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive a single dose of AG 920 or Proparacaine into one (study) eye.

Each dose of AG-920 or Proparacaine HCl will consist of two drops in the study eye. After the completion of dosing, subjects will undergo an eye exam, and the ability to conduct that eye exam will be documented. Investigational medicinal product (IMP) dosing will be performed by the study staff.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-pubescent with no childbearing potential
2. Capable of undergoing an eye exam
3. Subject's legally appointed and authorized representative willing to sign and date an informed consent form (ICF) and, where appropriate, the subject willing to sign an assent form prior to any study-related procedures being performed.
4. Parent/legal guardian and subject are willing and able to follow instructions and can be present for the required study visits and Follow-up Phone Call for the duration of the study.
5. Have a healthy, normal cornea.

Exclusion Criteria:

1. Have participated in an investigational study (drug or device) within the past 30 days.
2. Have a known contraindication to local anesthetics.
3. Children with known autism spectrum disorders or known to have heightened sensitivity.
4. Corneal pathology that would make the corneal sensitivity lower/higher or make the test hard to perform or interpret.
5. Have low visual acuity
6. Manifest nystagmus
7. Have had ocular surgery or general surgery within the past 45 days.
8. Have had an intravitreal injection in either eye within 14 days of randomization.
9. Have ocular surface disease.

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Uram, MD, Study Director — Medical Expert
Locations (1):
- American Genomics Site 2, McAllen, Texas, United States

REFERENCES:
- [Derived] Gonzalez VH, Uram M, Schupp A, Widmann M, Novack GD. AG-920 (Articaine) Ophthalmic Solution: A Masked, Active-Controlled Evaluation of Its Local Anesthetic Efficacy and Safety in Pediatric Patients. J Ocul Pharmacol Ther. 2024 Jun;40(5):293-296. doi: 10.1089/jop.2023.0187. Epub 2024 Apr 22. PMID 38647654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty (60) pediatric subjects were randomized and treated in a phase 1 unit between 6 April 2022 to 27 May 2022.
Period: Overall Study
Arm/Group | AG-920 | Proparacaine
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Four analysis populations were defined: Randomized Population, Safety Population, Intent-to-Treat (ITT) Population , Per-Protocol (PP) Population. The safety, ITT and PP populations included 60 subjects. Randomized Population completed Day 1. Safety Population are subjects who received at least one drop of the dose (2 drops). ITT subjects received at least one dose (2 drops) and PP population were all randomized subjects who completed the study treatment with no major protocol violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | AG-920 | Proparacaine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (3.1) | 6.3 (2.5) | 5.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Study Eye [Count of Participants; unit: Participants]
  Left Eye | 15 | 15 | 30
  Right Eye | 15 | 15 | 30
Color of Iris [Count of Participants; unit: Participants]
  Brown | 30 | 28 | 58
  Green | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants in Which an Eye Exam Was Able to be Performed
Description: Was the investigator was able to perform the eye examination without additional anesthesia
Time Frame: Two to four minutes following treatment (last drop) of IMP
Measure: Count of Participants; unit: Participants
Arm/Group | AG-920 | Proparacaine
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs will be summarized by treatment group using frequency and percent for each system, organ, class (SOC) and preferred term within each SOC. Summaries will be presented separately for ocular and non-ocular Adverse Events (AEs).
Time Frame: From randomization through study completion (up to 4 days following treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AG-920 | Proparacaine
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time the subject was consented until the subject's participation in the study was completed. If a subject had an ongoing AE at the time of study completion, the event was to be followed-up according to the site's standard of care and the subject provided appropriate medical care until the event resolved or stabilized.
Arm/Group | AG-920 | Proparacaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Language in clinical trial agreement states:

INVESTIGATIVE SITE, the Principal Investigator, and any other investigators understand and agree that the Study is a multi-center clinical study and that a multi- center publication may be prepared and published by the Sponsor. The INVESTIGATIVE SITE and its investigators will not, individually or together, present or publish any findings, data or results of the Study.

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT05325853/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT05325853/SAP_001.pdf